CLINICAL TRIAL: NCT02871271
Title: Open-Label Pilot Study to Evaluate the Tolerability and Benefit of IQP-AS-121 on Fatigue and Mental Alertness in Healthy Subjects
Brief Title: Tolerability and Benefit of IQP-AS-121 on Fatigue and Mental Alertness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped product production
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INQ/009416
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2016-07

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IQP-AS-121 (Experimental): To be taken once daily dosing of 1 tablet in the morning.
  Interventions: Dietary Supplement: IQP-AS-121

INTERVENTIONS:
Dietary Supplement: IQP-AS-121

SUMMARY:
The purpose of this study is to evaluate the tolerability and benefit of IQP-AS-121 on reducing fatigue and tiredness and to improve mental alertness.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian males and females, 21-55 years of age
2. Body mass index (BMI) 18.5-29.9 kg/m2
3. Generally in good health without clinically significant findings at screening
4. No chronic fatigue syndrome according to the Fukuda Centres for Disease Control and Prevention (CDC) criteria at screening
5. Subjective feeling of chronic stress and tiredness for 3-12 last months prior to screening
6. Screening Scale of Chronic Stress (SSCS) score >18
7. Fatigue Severity Scale score >4
8. ≤ 3 cups/portions of coffee and/or caffeine-containing food/beverages per day in the 3 last months prior to screening and during the study
9. Regular stable continuous level of daily activities
10. Regular sleep-wake cycle
11. Normal dietary habits according to investigator's judgement
12. ≤ moderate level of physical exercise
13. Readiness to comply with study procedures, in particular:

    * Consumption of the IP during the treatment period
    * Filling in all questionnaires
    * Keep habitual diet and level of physical exercise
14. No change in smoking habits during the study
15. Women of child-bearing potential only:

    1. negative pregnancy testing (ß-HCG in urine at screening)
    2. commitment to use reliable contraception methods during the entire study Participation is based upon written informed consent form (ICF) by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known sensitivity to any components of the IP
2. Any medical condition associated with tiredness (e.g. iron deficiency, hypotension etc.)
3. History and/or presence of clinically significant disease, which per investigator's judgement could interfere with the results of the study or the safety of the subject:

   1. Psychiatric diseases, e.g. depression, schizophrenia
   2. Eating disorders such as anorexia
   3. Untreated or non-stabilized metabolic diseases, e.g. diabetes mellitus
   4. Untreated or non-stabilized thyroid disorder
   5. Untreated or non-stabilized hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg)
   6. Significant gastrointestinal diseases
   7. Insomnia
   8. Known bleeding disorders such as haemophilia
   9. Any other known significant or serious condition / disease that renders subjects ineligible (e.g. history of malignancy within the past 5 years prior to screening, any clinically significant cardiovascular, renal, liver disease etc.)
4. Use of medication which in the investigator's judgement could interfere with the results of the study (e.g. psychoactive medication, statins, proton pump inhibitors, blood-pressure medications, antihistamines, antibiotics, diuretics) within the last 4 weeks prior to screening and during the study
5. Consumption of vitamins, nutritional supplements, supplementary balanced diet, mineral products which in the investigator's judgement could interfere with the results of the study within last 4 weeks prior to screening and during the study
6. Consumption of adaptogens (e.g. ginseng or Schisandra) or St. John's Wort within last 4 weeks prior to screening and during the study
7. Consumption of energy drinks during the study
8. Start of use of contraception medication during the last 3 months prior to screening and during the study
9. Use of anticoagulants such as warfarin
10. Clinically significant deviation of laboratory parameters and/or deviations > 2 x ULN (upper limit of normal) at screening
11. Recent or current significant stressors (e.g. active grieving)
12. Chronic pain
13. Chronic sleep deficiency (< 5 hours/night)
14. Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
15. Drug abuse
16. Participation in another study during the last 30 days prior to screening
17. Women of child-bearing potential: pregnant or breastfeeding
18. Any situation expected during the study causing acute high level of stress
19. Any other reason deemed suitable for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Estimated); Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in VAS-F parameter | 6 weeks
  Compared between timepoints week 6 versus baseline
  - To assess fatigue and energy with 18 items which possesses two subscales: fatigue (13 items) and energy (5 items).

SECONDARY OUTCOMES:
Change in Bond & Lader VAS parameter | 6 weeks
  Compared between timepoints week 6 versus baseline
  - To assess alertness, contentedness and calmness
Change in Number Connection Test | 6 weeks
  Compared between timepoints week 6 versus baseline
  - To assess visuo-spatial orientation and cognitive processing speed.
Change in FAIR-2 | 6 weeks
  Compared between timepoints week 6 versus baseline
  - To measure attention as an ability to concentrate
Change in SF-12 parameter | 6 weeks
  Compared between timepoints week 6 versus baseline
  - To measure the overall health status of a subject
Change in PSQ20 parameter | 6 weeks
  Compared between timepoints week 6 versus baseline
  - Contained 30 items as an instrument to assess subjectively experienced stress
Change in POMS-35 parameters | 6 weeks
  Compared between timepoints week 6 versus baseline
  - The POMS-65 comprises 65 adjectives, separated into 6 subscales: 1) depression-dejection, 2) tension-anxiety, 3) anger-hostility, 4) confusion bewilderment, 5) fatigue-inertia and 6) vigour-activity.
Global evaluation of benefit | 6 weeks
  Assessed by the subjects and investigator at the end of study
  - To evaluate benefit of IP
Adverse events | 6 weeks
  Assessed throughout the study
Global evaluation of tolerability | 6 weeks
  Assessed by the subjects and investigator at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack,, MD, PhD, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No